CLINICAL TRIAL: NCT04959214
Title: The Effect of Progressive Relaxation Exercises Applied to Nurses Working in the Intensive Care Unit on Sleep Quality and Fatigue Severity
Brief Title: The Effect Of Progressıve Relaxatıon Exercıses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seren (Other)
Responsible Party: Sponsor-Investigator, Seren, Master Student, Cukurova University
Organization: Cukurova University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10359740
Record Dates: First submitted 2021-06-29; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Sleep Disturbance; Fatigue
Keywords: Nurse; Progressive Relaxation; Sleep; Intensive Care; Fatigue
MeSH Terms: conditions — Parasomnias; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention: progressive relaxation exercise practice group (Experimental): intervention: progressive relaxation exercise practice group: A group of 30 intensive care nurses who will practice the progressive relaxation exercise at home 3 days a week for 1 month.
  Interventions: Behavioral: progressive relaxation egzersize
- control: uninterrupted group (No Intervention): control: A group of 30 intensive care nurses who did not intervene for 1 month

INTERVENTIONS:
Behavioral: progressive relaxation egzersize — Performing exercises in a quiet environment for 45 minutes with the Turkish Psychologists Association CD. Filling the PSQI and FSS before and 1 month after the application
  Arms: intervention: progressive relaxation exercise practice group

SUMMARY:
This study was conducted to evaluate the effect of progressive relaxation exercises applied to nurses working in the intensive care unit three times a week for 1 month on sleep quality and severity of fatigue. The research is a pretest-posttest randomized controlled study with an intervention control group.

DETAILED DESCRIPTION:
The Effect of Progressive Relaxation Exercises Applied to Nurses Working in The İntensive Care Unit on Sleep Quality and Fatique İntensity The study was planned to determine the effect of progressive relaxation exercises applied to nurses working in intensive care units on sleep quality and fatigue intensity.

The study will be conducted with a randomized controlled experimental research design in order to evaluate the effect of progressive relaxation exercises applied to nurses working in the intensive care unit on sleep quality and fatigue intensity. This randomized controlled study will be conducted on nurses working in Adana City Training and Research Hospital Intensive Care Unit. Nurses will be divided into 2 groups as experiment and control. It will be carried out on 60 people in total, 30 for the experimental group, 30 for the control group. Progressive relaxation exercises will be applied by nurses for 45 minutes, 3 days a week for an average of 1 month.

The data of the study will be collected after the purpose of the study is explained to the nurses and their verbal and written consents are obtained. In the collection of research data, the Personal Information Form prepared by the researchers and containing the introductory information of the nurses, the Pittsburgh Sleep Quality Index (Pittsburgh Sleep Quality Index Scale PSQI), the Fatigue Severity Scale for fatigue (FSS) will be collected from control and intervention groups through face-to-face interviews.

There are a limited number of studies showing the effects of progressive relaxation exercises applied to intensive care nurses on sleep quality and fatigue intensity in our country. With the study, the use of these exercise programs, which can be easily applied by nurses who work under heavy workloads in the intensive care environment, will increase, and it will be ensured that nurses work more fit and efficiently and are supported in terms of sleep fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Without a psychiatric diagnosis,
* Having a score of PUKI ≥5 and YŞÖ≥4,
* Nurses who volunteered to participate in the study were included in the research sample.

Exclusion Criteria:

* Experience of working in intensive care for less than 3 months,
* Using antidepressant, antihistamine, diuretic, hypnotic, benzodiazepine, antidepressant, anxiolytic and narcotic analgesics that affect sleep quality,
* Pregnant nurses were not included in the research sample.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
Post-application fatigue severity rate of nurses working in the intensive care unit | Scales are filled before starting the application and at the end of the application after 1 month.
  Fatigue severity scale The scale developed by Krup (1989) is a nine-item scale that evaluates the overall effect of fatigue on daily activities.In the scale, individuals are asked to rate the fatigue they have felt during the past week from 1 to 7. The total score is calculated by taking the average of nine items. The cut-off value for pathological fatigue was determined as 4 and above. The lower the total score, the less fatigue.
Decrease in sleep quality scale scores after the application | Scales are filled before starting the application and at the end of the application after 1 month.
  The Pittsburgh Sleep Quality Index (PUKI, PSQI) was developed in 1989 by Buysse et al. (Buysee et al, 1989) to evaluate sleep quality in the last month. The scale consists of a total of 24 questions, 19 of which were answered by the individual and five of them by the relatives of the individual.Each item score varies between "0" and "3", and the sum of the scores of the items in the seven components gives the scale score of 18.The total PUKI score ranges from 0 to 21. If this score is above 5, it indicates that the sleep quality of the individual is poor.

CONTACTS AND LOCATIONS:
Overall Officials: Songül Karadağ, Principal Investigator — Cukurova University
Locations (1):
- Cukurova University, Sarıçam, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Results of intervention and control group scales before and after administration (statistical analysis) Introductory characteristics of the participants and participant consent form
Supporting Information: SAP, ICF
Time Frame: Data is continuously available after publication
Access Criteria: Data can be shared publicly
URL: https://tez.yok.gov.tr/UlusalTezMerkezi/